CLINICAL TRIAL: NCT06258616
Title: Fluid Administration and Fluid Accumulation in the Intensive Care Unit (FLUID-ICU) - an International Inception Cohort Study
Brief Title: Fluid Administration and Fluid Accumulation in the Intensive Care Unit
Acronym: FLUID-ICU
Status: Recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: FLUID-ICU
Record Dates: First submitted 2024-01-22; First posted 2024-02-14 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Fluid Accumulation; Fluid Therapy; Fluid Overload
Keywords: Fluid Overload; Fluid Accumulation; Fluid Administration
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this international inception cohort study is to describe fluid administration during admittance to the intensive care unit (ICU), and provide contemporary epidemiological data on fluid accumulation, risk factors, management and outcome in critically ill adult patients.

DETAILED DESCRIPTION:
Background: Fluid accumulation is associated with adverse outcome in ICU patients, however, assessment of fluid status is often difficult and no established definition and consistent detection method exists. Former research has primarily focused on the use of resuscitation fluid, but a substantial amount of fluid is administered throughout the entire ICU stay and this fluid may be a clinically relevant source of fluid accumulation.

Objectives: To describe fluid administration practices during the entire ICU stay, and provide contemporary epidemiological data on fluid accumulation, fluid removal, risk factors and association with patient outcomes from a worldwide perspective.

Study design: International inception cohort study. Patients will be included during a 14-day inception period to be chosen by each participating site.

Population: Critically ill adult patients (≥ 18 years) with acute admission to the ICU.

Intervention: None. Only routinely available data will be collected.

Study duration: Patients are followed daily until ICU discharge or death for a maximum of 28 days. Follow-up is performed 90 days after ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Acute admission to the ICU during the 14-day inception period.
* Adults (≥ 18 years).

Exclusion Criteria:

* Patients previously included in the FLUID-ICU study.
* Patients with major burns (≥ 10% of body surface)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the participating ICUs during the 14-inception period.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The number of patients with fluid accumulation. | From ICU admission to discharge (with a maximum of 28 days).
  The presence of fluid accumulation is defined as the best clinical estimate made by the study investigators, using medical records and the treating team's clinical assessment, and one or more of the following parameters: Cumulative fluid balance, daily fluid balance, changes in body weight, and/or clinical signs of fluid accumulation (e.g. peripheral oedema, pulmonary oedema, congestion on chest X-ray or lung ultrasound).

SECONDARY OUTCOMES:
Number of patients with fluid accumulation upon ICU admission (baseline). | On the first day of ICU admission (Day 1).
  Defined as the number of patients with fluid accumulation upon ICU admission or equal to the time of ICU assessed by study investigators using cumulative fluid balance, daily fluid balance, changes in body weight and clinical signs of fluid accumulation.
Number of patients developing fluid accumulation during the ICU stay. | 28 days
  Defined as the number of patients developing fluid accumulation during ICU stay (one or more episodes) but no pre-existing fluid accumulation upon ICU admission (baseline form).
Number of days with fluid accumulation during the ICU stay. | 28 days
  Defined as the median number of days with fluid accumulation in patient with fluid accumulation at baseline and/or during ICU stay at day 28 after ICU admission.
Number of patients being treated with 'active fluid removal' (use of diuretics, or renal replacement therapy). | 28 days
  Defined as patients that receive treatment with any type of diuretics or renal replacement therapy.
Days alive without use of life-support within 28 days from ICU admission. | 28 days
  Days alive without use of life-support (continuous infusion of vasopressors/inotropes, invasive mechanical ventilation or renal replacement therapy).
Days alive and out of hospital within 90 days from ICU admission. | 90 days
  Total number of days alive and out of hospital within 90 days from ICU admission,
Mortality within 90 days from ICU admission. | 90 days
  Death from all causes.

OTHER OUTCOMES:
The volume (mL) of fluid administered day 1-7 and after 28 days in the following categories: Resuscitation fluid, maintenance-replacement fluid, fluid creep, nutrition, blood products. | Day 1-7 and after 28 days.
  Definition: the median volume of all fluid in millilitres (mL) administered during ICU admission categorized by indication (resuscitation, maintenance-replacement, fluid creep, nutrition, blood products) reported on day 1, 2, 3, 4, 5, 6, 7 and 28 days after ICU admission.
Fluid balance (mL) during ICU stay on day 1-7 and 28 days after ICU admission | Day 1-7 and after 28 days
  Definition: The sum of all daily fluid inputs minus all daily fluid outputs reported on day 1, 2, 3, 4, 5, 6, 7 and 28 days after ICU admission in mL (median).
Cumulative fluid balance (mL) day 1-7 and 28 days after ICU admission | Day 1-7 and after 28 days.
  Definition: Cumulative fluid balance will be calculated as the sum of all fluid input minus all fluid output reported on day 1, 2, 3, 4, 5, 6, 7 and 28 days after ICU admission in mL (median).

CONTACTS AND LOCATIONS:
Locations (21):
- Denmark (11):
  - Deparment of Intensive care, Nordsjællands hospital, Hillerød, Hillerød
  - Department of Intensive Care, Sygehus Sønderjylland Aabenraa, Aabenraa
  - Departmen of Intensive Care, Aalborg
  - Department of Intensive Care, University hospital Aarhus, Aarhus
  - Department of Intensive Care, Rigshospitalet 4131, Copenhagen
  - Department of Intensive Care, Bispebjerg, Copenhagen
  - Department of Intensive Care, Herlev Hospital, Herlev
  - Department of Intensive Care, Regionshospital Gødstrup, Herning
  - Department of Intensive Care, Zealand University hospital, Køge
  - Department of Intensive Care, Regionshospitalet Randers, Randers
  - Department of Intensive Care, University Hospital Zealand, Roskilde, Roskilde
- Department of Intensive Care, Tampere University Hospital, Tampere, Finland
- Department of Intensive Care, Landspitali National University Hospital of Iceland, Reykjavik, Iceland
- Department of Anaesthesiology, Critical Care and Pain Tata Memorial Hospital, Mumbai., Mumbai, India
- Department of Anaesthesia and Critical Care Vilnuis University Hospital Santariskiu Cinics, Vilnuis, Vilnius, Lithuania
- Department of Intensive Care Wellington Hospital (CCDHB), Newton, Wellington, Wellington, New Zealand
- Department of Intensive Care, Stavanger University Hospital, Stavanger, Norway
- Hospital Clinic of Barcelona, Barcelona, Spain
- Helsingborg Hospital, Helsingborg, Sweden
- Department of Intensive Care, Inselspital, Bern, Switzerland
- General Adult Intensive Care Unit, Critical Care Directorate University Hospital of Wales, Cardiff, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No